CLINICAL TRIAL: NCT01009008
Title: Patient Activated Controlled Expansion (PACE) for Breast Reconstruction Utilizing Controlled CO2 Inflation
Brief Title: Patient Activated Controlled Expansion (PACE) Trial
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AirXpanders, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-0001
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer; Mastectomy; Breast Reconstruction
Keywords: cancer; breast cancer; mastectomy; breast reconstruction; reconstruction; tissue expansion; two-stage breast reconstruction; tissue expander; AeroForm; AirXpander
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Post-mastectomy (Experimental): Post-mastectomy patients undergoing expander reconstruction
  Interventions: Device: Patient Activated Controlled Expansion Device

INTERVENTIONS:
Device: Patient Activated Controlled Expansion Device — Patient activated controlled expansion for post-mastectomy breast reconstruction

SUMMARY:
The purpose of this study is to determine whether a patient controlled tissue expander can improve the results and patient experience in breast reconstruction. The study hypothesis is that patient controlled expansion will lead to rapid and more comfortable outcomes than historical precedents.

DETAILED DESCRIPTION:
Title: Patient Activated Controlled Expansion (PACE) for Breast Reconstruction Utilizing Controlled CO2 Inflation

Design: Prospective, open-label, single-arm, feasibility trial Purpose: To evaluate the AirXpanders tissue expander in patients undergoing breast reconstruction surgery following mastectomy.

Enrollment: This feasibility trial will enroll up to 10 patients. Following enrollment of the first 5 patients, the sponsor will determine if additional subjects will be recruited to further evaluate treatment outcome.

Clinical Sites: Up to 3 sites and 3 surgeons will participate in this study. The surgeon(s) should have the necessary qualifications and sufficient experience (minimum of 12 breast tissue expanders placed per year) to participate in the trial.

Duration of Patient Participation: Eligible patients will be enrolled over approximately 2 months.

Patients will be instructed on the tissue expansion protocol pre-operatively and undergo post-operative clinical follow-up on a weekly basis or more frequently if deemed necessary by the treating surgeon.

Each patient will be followed through removal of the tissue expander.

Study Population:

The study population will consist of up to 10 patients. Eligible patients are females between the ages of 18 and 65 years who are planning to undergo breast reconstruction surgery following mastectomy. Eligible patients must be able to provide informed consent and understand protocol components.

ELIGIBILITY:
Inclusion Criteria:

1. Female between the ages of 18 and 65 years.
2. Planned breast reconstruction surgery post-mastectomy.
3. Able to provide informed consent.
4. Able to understand protocol components.

Exclusion Criteria:

1. Tissue at the intended expansion site is determined unsuitable by the surgeon (i.e., infection, compromised vascularity, history of compromised wound healing, mastectomy skin flaps of questionable viability, excessively tight skin envelope, previous radiation treatment, active ulceration)
2. Residual gross tumor at the intended expansion site
3. History of or planned adjuvant radiation therapy
4. Co-morbid condition determined by the surgeon to pose unduly high risk of surgical and/or postoperative complications.
5. Obesity with BMI of 30 or above
6. Current smoker
7. Psychologically unsuitable patient
8. Patient unable to understand the protocol for tissue expansion
9. Planned flight or assent to altitude exceeding 1000 meters above baseline during the expansion period.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Expansion to and maintenance of clinically desired breast volume (not exceeding implant maximum) until permanent implant placement or 6 months (whichever comes first) unless prohibited by a non-device related failure. | 6 months

SECONDARY OUTCOMES:
Safety as evidenced by a low incidence of device-related adverse events. | 6 months
Time required to achieve desired expansion results. | 6 months
Overall patient treatment satisfaction. | 6 months
Overall surgeon treatment satisfaction. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Connell, M.D., Principal Investigator
Locations (1):
- The Mount Hospital, Perth, Western Australia, Australia

REFERENCES:
- [Derived] Connell TF. Patient-activated controlled expansion for breast reconstruction using controlled carbon dioxide inflation: confirmation of a feasibility study. Plast Reconstr Surg. 2014 Oct;134(4):503e-511e. doi: 10.1097/PRS.0000000000000551. PMID 25357043
- [Derived] Connell AF. Patient-activated controlled expansion for breast reconstruction with controlled carbon dioxide inflation: a feasibility study. Plast Reconstr Surg. 2011 Oct;128(4):848-852. doi: 10.1097/PRS.0b013e3182268b80. PMID 21921761